CLINICAL TRIAL: NCT05125042
Title: A Randomized Control Study of Catgut Embedding in Acupoint on Treating Persistent Atrial Fibrillation After Catheter Ablation: a Chinese Registry Study.
Brief Title: Catgut Embedding in Acupoints on Treating Persistent Atrial Fibrillation After Catheter Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, deputy director of cardiology department of Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAF
Record Dates: First submitted 2021-11-17; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation after catheter ablation; catgut embedding in acupoints
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Amiodarone hydrochloride tablet + acupoint catgut embedding of Neiguan and Zusanli
  Interventions: Procedure: Amiodarone hydrochloride tablet + acupoint catgut embedding; Drug: Amiodarone hydrochloride tablet
- group B (Active Comparator): Amiodarone hydrochloride tablet
  Interventions: Procedure: Amiodarone hydrochloride tablet + acupoint catgut embedding; Drug: Amiodarone hydrochloride tablet

INTERVENTIONS:
Procedure: Amiodarone hydrochloride tablet + acupoint catgut embedding — Patients with persistent AF after undergoing catheter ablation take receive acupoint catgut embedding in Neiguan and Zusanli twice after and one month after surgery combined with amiodarone hydrochloride tablets 200mg bid, 1 month; 200mg qd,maintained to 3 months.All patients, who had no signs of recurrence three months after surgery, stopped taking medication.
Drug: Amiodarone hydrochloride tablet — Patients with persistent AF after undergoing catheter ablation only take amiodarone hydrochloride tablets 200mg bid, 1 month; 200mg qd,maintained to 3 months.All patients, who had no signs of recurrence three months after surgery, stopped taking medication.

SUMMARY:
This is a multi-center, 2-arm, assessor and statistician blinded, pilot randomized controlled trial, to evaluate the effect of catgut embedding in acupoints of Neiguan and Zusanli in reducing early recurrence and improving long-term prognosis in patients with persistent AF after CA..

DETAILED DESCRIPTION:
This multi-center, 2-arm, assessor and statistician blinded, pilot randomized controlled trial will be conducted at two centers in China: Shanghai Chest Hospital; The Second Affiliated Hospital of Shandong University of traditional Chinese Medicine. Patients with persistent atrial fibrillation after catheter ablation are 1:1 randomized into group A (amiodarone hydrochloride tablet + acupoint catgut embedding), group B (amiodarone hydrochloride tablet). ECG, inflammatory cytokines,AFEQT scale and other indicators are analyzed the effect of catgut embedding in acupoints of Neiguan and Zusanli in reducing early recurrence and improving long-term prognosis in patients with persistent AF after CA.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18 and 80 years old; 2. Persistent AF（lasting no more than 3 years）after catheter ablation; 3. No acupuncture treatment within the previous 6 months.

Exclusion Criteria:

* 1. A history of allergy to acupuncture or amiodarone; 2. Severe heart failure (New York Heart Association（NYHA）class III or IV); 3. Echocardiographic parameters: left ventricular ejection fraction < 40%, left atrium diameter > 5.0cm; 4. Severe lung, liver, kidney disease or other serious primary diseases; 5. Skin allergy to ECG monitoring electrode patch. 6. The estimated life expectancy of < 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation (AF)/atrial flutter (AFL)/atrial tachycardia (AT) recurrence rate | 12 months after ablation
  at 12 months (AF/AFL/AT recurrence is defined as presence of documented AF/AFL/AT episodes of 30 seconds or longer duration).

SECONDARY OUTCOMES:
Postoperative AF recurrence rate | up to 12 months after ablation
  AF recurrence is defined as presence of documented AF episodes of 30 seconds or longer duration
TCM symptom score scale | up to 12 months after ablation
Inflammatory index | up to 12 months after ablation
AF-specific Atrial Fibrillation Effect on QualiTy-of-life Scale | up to 12 months after ablation